CLINICAL TRIAL: NCT04013984
Title: The Effect of Acupuncture on in Vitro Fertilization/ Intracytoplasmic Sperm Injection Embryo Transfer (IVF/ICSI-ET) Outcomes in Patients With Poor Ovarian Response Diagnosis: A Randomized Controlled Trial
Brief Title: Acupuncture for Treatment of Patients With Poor Ovarian Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POR-accupuncure
Record Dates: First submitted 2019-04-08; First posted 2019-07-10 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Poor Ovarian Response; Accupuncture

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Accupuncture (Experimental): Acupuncture twice a week during the preceding cycle and the ovarian stimulation by "GnRH agonist stopped protocol".
  Interventions: Other: Accupuncture
- Non-accupuncture (No Intervention): Ovarian stimulation by" GnRH agonist stopped protocol" without intervention.

INTERVENTIONS:
Other: Accupuncture — In experimental groups (A), acupuncture will be applied for 30 minutes in each session and will be started from the month prior to onset of ovarian stimulation (two sessions of a weekly), and during the ovarian stimulation cycle (two sessions of a weekly), totally 7 acupuncture sessions will be carried out. Acupuncture will be performed using sterile needle on specific points (CV 3 (Zhongji), CV 4 (Guanyuan), ST 25 (Tianshu), ST 28 (Shuidao), ST 29 (Guilai), and LR 3 (Taichong), BL 23 (Shenshu), BL 32 (Ciliao), GV 20 (Baihui), GV 24 (Shenting), GB 13 (Benshen), ST 36 (Zusanli), SP 6 Sanyinjiao), SP 8, SP 10 and KI 3 (Taixi)). The needles were inserted to a depth of 15-30 mm, depending on the region of the body. No sham acupuncture is considered in the control group for ethical and practical reasons
  Arms: Accupuncture

SUMMARY:
This prospective randomized controlled trial is designed to investigate the effect of acupuncture on IVF/ICSI outcome in women with poor ovarian response. The study population consisted of all infertile women with a previous poor ovarian response who will undergo IVF/ICSI in Reproductive Biomedicine Research Center, Royan institute, Tehran Iran. To minimize the effect of ovarian stimulation protocol, a stratified randomization method according to ovarian stimulation protocols (GnRH agonist stopped and GnRH antagonist) is used.

DETAILED DESCRIPTION:
Poor ovarian response (POR) is a challenging issue in assisted reproduction treatment. Different controlled ovarian hyperstimulation protocols and strategies have been used in this group of women to improve reproductive outcome, but the success rate still remains low. The aim of this study was to determine the effect of acupuncture during ovulation induction on the results of IVF / ICSI cycles in patients with POR diagnosis. The study was approved by the institutional review board. Written, informed consent will be obtained from each participant. Infertile women with a diagnosis of POR, who undergoing the IVF / ICSI cycle are assigned to four groups by stratified randomization method according to ovarian stimulation protocol. Before the starting the treatment cycle, patients will be randomized with sealed randomization envelopes. The random allocation is concealed from the physician performing the IVF/ICSI treatment cycle. All patients will receive acupuncture by the same physician (Dr.Salimi). In experimental groups (A), acupuncture will be applied for 30 minutes in each session and will be started from the month prior to onset of ovarian stimulation (two sessions of a weekly), and during the ovarian stimulation cycle (two sessions of a weekly), totally 7 acupuncture sessions will be carried out. Acupuncture will be performed using sterile needle on specific points (CV 3 (Zhongji), CV 4 (Guanyuan), ST 25 (Tianshu), ST 28 (Shuidao), ST 29 (Guilai), and LR 3 (Taichong), BL 23 (Shenshu), BL 32 (Ciliao), GV 20 (Baihui), GV 24 (Shenting), GB 13 (Benshen), ST 36 (Zusanli), SP 6 Sanyinjiao), SP 8, SP 10 and KI 3 (Taixi)). The needles were inserted to a depth of 15-30 mm, depending on the region of the body. No sham acupuncture is considered in the control group for ethical and practical reasons. There is no intervention in the control groups (B).

Controlled ovarian stimulation for patients in both groups will be performed according the long stopped protocol. GnRH agonist (Buserelin, 0.5 mg), beginning on day 18 of the previous cycle will be used for down regulation and then will be stopped on the starting ovarian stimulation. Ovarian stimulation will be done with recombinant FSH and hMG (225 IU recombinant FSH (Gonal-F®; Serono Laboratories Ltd., Geneva, Switzerland) and 75 IU hMG (Menopur®; Ferring). The doses of gonadotropins were adjusted as ovarian response in the ultrasound monitoring. Ovulation was triggered with hCG (10,000 IU) when at least three follicles have a diameter of 18 mm with an adequate serum E2 concentration.

In both group, transvaginal oocyte retrieval will be performed under ultrasound guidance 32-34 hours after hCG administration. Intracytoplasmic sperm injection will be performed for all metaphase II oocytes. Embryo transfer will be done under ultrasound guidance on day 3 for all patients.

Primary consequences in this study are the total number of retrieved and MII oocytes and quality of the obtained embryos. Secondary outcomes are implantation and clinical pregnancy rates that confirmed by vaginal ultrasound (pregnancy sac and embryonic heart activity). The IVF/ICSI outcomes are compared in four groups. Data collection will be performed by using questionnaire to be filled as per the available records and laboratory results. Data analysis will be done through descriptive and perceptive statistical methods by using SPSS software version 20 for windows.

ELIGIBILITY:
Inclusion Criteria:

1- Diagnosis of Poor ovarian response (POR), according to POSSEIDON group criteria (Group 3) Young patients (<35 years) with poor ovarian reserve prestimulation parameters (AFC <5, AMH<1.2 ng/mL).

Exclusion Criteria:

1. Premature ovarian failure diagnosis.
2. Endometriosis grade III or IV.
3. Any contraindications to ovarian stimulation treatment.
4. Uterine infertility factor.
5. Previous history of ovarian surgery.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Total number of retrieved oocytes | Day of oocyte pick-up, 34-36 hours after hCG administration (approximately Stimulation Day 10)
  At the point of ovum pick-up, we can count total number of retrieved oocytes. Therefore, in one hour after ovum pick-up, outcome measurement will be possible.
Oocyte maturity | Day of oocyte pick-up, 34-36 hours after hCG administration (approximately Stimulation Day 10)
  At the point of ovum pick-up, we can count how many mature or immature oocytes were retrieved. Therefore, in one hour after ovum pick-up, outcome measurement will be possible.
Quality of obtained embryos | 3 days after IVF/ICSI procedure
  Embryo grade assessed under invert microscope 3 days after intracytoplasmic sperm injection procedure [ Time Frame: 3 days after intracytoplasmic sperm injection procedure ] Embryo grade assessed under invert microscope 3 days after intracytoplasmic sperm injection procedure.The quality of embryos was graded from 1 to 3 under inverted microscope 3 days after intracytoplasmic sperm injection procedure. Embryos with even-sized blastomers and/or <5% fragments were classified as Grade 1 (good quality). Grade 2 embryos (moderate quality) had blastomeres with slightly-moderate size differences and/or 5-50% fragments. Grade 3 embryos (poor quality) had markedly different-sized blastomers and/or >50% fragments.

SECONDARY OUTCOMES:
Implantation rate | 4 weeks after embryo transfer
  The ratio of total number of observed gestational sacs to total number of transferred embryos.
Clinical pregnancy rate | 4-6 weeks after embryo transfer
  The observation of gestational sac with heart beat by using trans-vaginal ulterasound

CONTACTS AND LOCATIONS:
Locations (1):
- Royan Institute, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No
We can share the results of study, after the publish the manuscript.